CLINICAL TRIAL: NCT05359978
Title: Occupational Therapy Intervention for Alzheimer's Disease Patients. An International Comparison in Spain and Italy.
Brief Title: Treatment in Occupational Therapy With Significant Activities to Improve Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Burgos (Other)
Responsible Party: Principal Investigator, OLALLA SAIZ VAZQUEZ, Graduado en Terapia Ocupacional, Universidad de Burgos
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Prevention
Other Study IDs: UBurgos2
Record Dates: First submitted 2022-04-20; First posted 2022-05-04 (Actual); Last update posted 2022-05-16 (Actual); Status verified 2022-05

CONDITIONS: Dementia
Keywords: Occupational Therapy; Dementia; Significance activities; No-pharmacological treatment
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Intervention Model Description: It's a pretest-posttest non-equivalent control group experimental design study comparing two cohorts of patient with different types of dementia
Who Masked: Participant
Masking Description: Approximately 250 patients will be screened to achieve 240 participants, divided in two cohorts (120 each), furthermore each cohorts was divided in other two groups (experimental group (60 each) and control group (60 each) the first one followed up by private centres in Spain endowed with Occupational Therapy and the second by public centres in the region of Modena
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cards (Experimental): participants received 2 days at week during 30 minutes
  Interventions: Behavioral: To with significance activities
- significance activities (Experimental): participants received 2 days a week during 30 minutes
  Interventions: Behavioral: To with significance activities

INTERVENTIONS:
Behavioral: To with significance activities — activities with purpose with people who are diagnosed of dementia 2 days at week during 30 minutes

SUMMARY:
We followed a pretest-posttest non-equivalent control group experimental design study comparing two cohorts of patient with different types of dementia.

Approximately 250 patients will be screened to achieve 240 participants, divided in two cohorts (120 each), furthermore each cohorts was divided in other two groups (experimental group (60 each) and control group (60 each) the first one followed up by private centres in Spain endowed with Occupational Therapy and the second by public centres in the region of Modena.

DETAILED DESCRIPTION:
The course of dementia goes through different stages and during the moderate and advanced stages cognitive decline and functional deterioration are frequently accompanied by the so-called behavioural and psychological symptoms of dementia (BPSD), that put severe stress on the persons with dementia (PwD), on their families and on the health system. Worldwide consensus guidelines recommend non-pharmacological approaches to be first line.

The occupational therapist studies human activity as a therapeutic resource to prevent and treat physical and/or psychosocial difficulties, in order to improve the person's quality of life.

Subjects were not randomly assigned to different treatment groups (control group and experimental group); instead, consecutive sampling was chosen by assigning subjects based on an odd-and-even-numbered technique (odd subjects were assigned to the control group and even subjects to the experimental group). Both groups presented the same pathological, cultural, and sexual characteristics, and belonged to the same age group.

ELIGIBILITY:
Inclusion Criteria:

* a diagnosis of primary dementia (DSM V)
* a MMSE score ≤ 24
* a NPI global score ≥ 32/144
* a treatment with significance activities in Occupational Therapy
* live in a nursing home

Exclusion Criteria:

* presence of uncontrolled medical disease potentially contributing to the cognitive decline and BPSD

  * concomitant psychiatric disorders or chronic alcoholism
  * concomitant diseases severe enough to reduce life expectancy < 6 months

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 240 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-03-20 (Actual); Study Completion 2022-04-20 (Actual)

PRIMARY OUTCOMES:
Tinetti | 2 days
  - The Tinetti test has been recommended and widely used in the elderly to assess mobility, balance and gait, and predict falls. Different versions can be found. A systematic literature search identified 37 publications on the Tinetti test and falls.
CDR | 2 days
  - The Clinical Dementia Rating (CDR) has demonstrated high validity and reliability for this purpose, but it requires a considerable amount of data to be collected both from the patient and from an informant.
MMSE | 2 days
  - The MMSE fulfilled its original goal of providing a brief screening test that quantitatively assesses the severity of cognitive impairment and documents cognitive changes occurring over time
NPI | 2 days
  - The NPI-Q Spanish version offers the possibility to use a reliable and brief instrument that can be used as a screening in the evaluation of neuropsychiatric symptoms in dementia and associated caregiver distress
Barthel | 2 days
  - Evidence suggests that (Barthel Index) BI is a valid measure of activities of daily living; sensitivity to change is limited at extremes of disability (floor and ceiling effects), and reliability of standard BI assessment is acceptable

CONTACTS AND LOCATIONS:
Locations (1):
- Olalla Saiz Vazquez, Burgos, Spain